CLINICAL TRIAL: NCT00093821
Title: A Multicenter Phase I Trial of 17-N-allylamino-17-demethoxy Geldanamycin (17-AAG, NSC #330507) in Patients With Recurrent/Refractory Pediatric Solid Tumors (Ewing's Sarcoma, Desmoplastic Small Round Cell Tumor, Osteosarcoma, Neuroblastoma, and Rhabdomyosarcoma) and Leukemia
Brief Title: Tanespimycin in Treating Young Patients With Recurrent or Refractory Leukemia or Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01456; 04-069; POETIC-MSKCC-04069; CDR0000391010; NCI-6323; MSKCC-04069; U01CA069856 (NIH)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Childhood Chronic Myelogenous Leukemia; Childhood Desmoplastic Small Round Cell Tumor; Disseminated Neuroblastoma; Metastatic Childhood Soft Tissue Sarcoma; Metastatic Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Metastatic Osteosarcoma; Previously Treated Childhood Rhabdomyosarcoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Neuroblastoma; Recurrent Osteosarcoma
MeSH Terms: conditions — Desmoplastic Small Round Cell Tumor; Neuroectodermal Tumors, Primitive, Peripheral; Osteosarcoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neuroblastoma | interventions — tanespimycin

ARMS (1):
- Treatment (tanespimycin) (Experimental): Patients receive tanespimycin IV over 2-6 hours on days 1, 4, 8, and 11 (for patients with solid tumors) OR days 1, 4, 8, 11, 15, and 18 (for patients with leukemia). Courses for all patients repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of tanespimycin until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 15 patients are treated at the MTD.
  Interventions: Drug: tanespimycin; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of tanespimycin in treating young patients with recurrent or refractory leukemia or selected solid tumors. Drugs used in chemotherapy, such as tanespimycin, work in different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose-limiting toxicity and maximum tolerated dose (MTD) of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) in pediatric patients with recurrent or refractory leukemia or selected solid tumors.

II. Determine the levels of key proteins known to influence cancer cell survival and proliferation in patients treated with this drug at the MTD.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics of this drug in these patients. II. Evaluate effects of genetic polymorphisms known to alter the activity of enzymes involved in the metabolism of this drug.

III. Correlate the alteration of fludeoxyglucose F18 accumulation with tumor response in patients treated with this drug.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to diagnosis (leukemia vs solid tumor).

Patients receive tanespimycin IV over 2-6 hours on days 1, 4, 8, and 11 (for patients with solid tumors) OR days 1, 4, 8, 11, 15, and 18 (for patients with leukemia). Courses for all patients repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of tanespimycin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 15 patients are treated at the MTD.

Patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of 1 of the following malignancies:

  * Leukemia

    * Lymphoid, myeloid, or mixed lineage
    * Relapsed (in second or greater relapse) or refractory disease, confirmed by 1 of the following:

      * Bone marrow relapse, defined as either M3 bone marrow (> 25% blasts in the bone marrow aspirate) OR M2 bone marrow (5-25% blasts in the bone marrow aspirate) at any time after complete remission is attained
      * CNS relapse, defined as at least 5 WBC/mL by cytospin of any cerebrospinal fluid (CSF) specimen OR less than 5 WBC/mL by cytospin of 2 consecutive CSF specimens obtained >= 4 weeks apart and having definitive confirmation that blasts are derived from the original leukemic clone by molecular cytogenetics, multiparameter flow cytometry, or immunostaining of >= 2 antigens
    * Patients with underlying chronic myeloid leukemia must have > 25% blasts in the bone marrow aspirate
    * Patients with M3 bone marrow AND extramedullary sites of disease, other than leptomeningeal disease, are eligible
  * Solid tumor

    * One of the following tumor types:

      * Neuroblastoma
      * Ewing's sarcoma
      * Osteosarcoma
      * Desmoplastic small round cell tumor
      * Rhabdomyosarcoma
    * Progressed after prior standard therapy OR no effective standard therapy exists
    * Measurable or nonmeasurable disease
* No known brain metastases
* No active leptomeningeal leukemia, defined by the following criteria:

  * WBC > 5/mm^3 in cerebrospinal fluid (CSF)
  * Unequivocal confirmation of leukemic blasts in CSF by cell morphology
* No symptomatic CNS disease (e.g., cranial nerve abnormalities) without cytologic abnormality in CSF
* Performance status - Karnofsky 70-100% (for patients > 10 years of age)
* Performance status - Lansky 70-100% (for patients =< 10 years of age)
* More than 8 weeks
* Absolute neutrophil count >= 750/mm^3
* Platelet count >= 75,000/mm^3 (transfusion independent)
* Hemoglobin >= 8.5 g/dL (transfusion allowed)
* Bilirubin < 1.5 mg/dL
* ALT and AST =< 2.5 times upper limit of normal (ULN)
* INR =< 1.5 times ULN
* Albumin > 2.0 g/dL
* Creatinine =< 1.5 times ULN for age
* Creatinine clearance or radioisotope glomerular filtration rate > 60 mL/min
* Ejection fraction >= 50%
* Shortening fraction >= 28%
* QTc < 450 msec for men (470 msec for women)

  * No congenital long QT syndrome
* LVEF > 40% by MUGA
* No symptomatic congestive heart failure
* No cardiac arrhythmia
* No New York Heart Association class III or IV heart failure
* No myocardial infarction within the past year
* No uncontrolled dysrhythmias
* No poorly controlled angina
* More than 12 months since active ischemic heart disease
* No history of serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation >= 3 beats in a row)
* No left bundle branch block
* No other significant cardiac disease
* No pulmonary fibrosis by radiography
* No ongoing or active bacterial or fungal infection
* No other uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No history of serious allergic reaction attributed to eggs or dimethyl sulfoxide
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Recovered from all immunotherapy
* At least 6 months since prior allogeneic stem cell transplantation
* At least 3 months since prior autologous stem cell transplantation
* At least 2 weeks since prior biologic agents (e.g., monoclonal antibodies)
* At least 1 week since prior filgrastim (G-CSF) or sargramostim (GM-CSF)
* Recovered from all prior chemotherapy
* At least 2 weeks since prior chemotherapy (for patients with leukemia only)
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) (for patients with solid tumors)
* No prior oxaliplatin
* No concurrent corticosteroids except for the treatment of adrenal crises in patients with suppressed hypothalamic-pituitary-adrenal axis response OR for treatment of allergic reactions to medications or blood products
* Recovered from all prior radiotherapy
* At least 6 months since prior radiotherapy to >= 50% of the pelvis
* At least 6 months since prior radiotherapy to substantial bone marrow, including total body irradiation
* At least 4 weeks since prior local (small port) radiotherapy
* No prior radiotherapy to the heart
* At least 1 week since prior retinoids
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent medication to control arrhythmias
* No concurrent medications that prolong or may prolong QTc interval
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2004-09; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
MTD, defined as the highest dose level with an observed incidence of DLT in no more than 1 out of 6 patients treated at a particular dose level | 21 days

SECONDARY OUTCOMES:
Change in Hsp90 client protein levels in relation to dose of tanespimycin | Baseline to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Trippett, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States